CLINICAL TRIAL: NCT02316366
Title: Clinical Impact of Warmed Intravenous Saline in Sickle Cell Patients With Vaso-Occlusive Episodes
Brief Title: The Use of Warmed Saline in Vaso-occlusive Episodes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Renee Quarrie, Attending, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB12-00295
Record Dates: First submitted 2014-12-10; First posted 2014-12-12 (Estimated); Results first posted 2015-08-31 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Sickle Cell Disease; Sickle Cell Crisis
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Warm fluid (Experimental): Patients in this arm of the study receive intravenous saline warmed to 37.5 degrees Celsius by Astoflo Plus fluid warmer
  Interventions: Device: Astoflo Plus fluid warmer
- Room temperature Fluid (No Intervention): Patients receive intravenous saline at room temperature (22-24 degrees Celsius)

INTERVENTIONS:
Device: Astoflo Plus fluid warmer — A fluid warmer (the Astoflo Plus warmer) was used to warm fluid to body temperature 37.5 degrees Celsius
  Arms: Warm fluid

SUMMARY:
The purpose of this study is to determine if warming the intravenous (IV) fluid given to patients with Sickle Cell Disease who are experiencing painful episodes known as Vaso-Occlusive Episodes; will decrease rates of hospital admission, decrease amounts of IV pain medications given, improve pain and improve global comfort.

DETAILED DESCRIPTION:
Vaso-occlusive crisis (VOC) is a common painful complication of Sickle Cell Disease and is the primary reason that these patients seek medical care in the acute care setting. This complication arises when blood vessels are obstructed by sickled red blood cells resulting in ischemic injury.

The standard management of these painful episodes comprises the administration of opioid analgesics, the infusion of intravenous (IV) fluids at room temperature and rest. These episodes often last five to seven days and many patients require inpatient management for continued administration of intravenous analgesics.

The public health impact of the disease is large as admissions frequently result in school or work absences and can be financially and emotionally taxing.

It is well established that exposure to cold precipitates VOC. For this reason, management of the pain of VOC in some centers includes the use of warming blankets as an adjunct for pain relief. It is conceptually appealing to conjecture that warm fluids might have similar salutary effects on VOC. This conjecture is bolstered by the physiologic effect of temperature on vascular tone. Specifically, it is well established that cold temperatures cause vasoconstriction whereas warm temperatures cause vasodilation. We expect that warmed fluids will similarly induce vasodilation, improving blood flow to vaso-occluded ischemic areas.

ELIGIBILITY:
Inclusion Criteria:

* Vaso-occlusive Episode defined as a pain rating of 3 or above on the Wong-Baker FACES score in a child with an established diagnosis of sickle cell disease (SS, SC or S β Thalassemia)
* 4-21 years of age

Exclusion Criteria:

* fever (temperature greater than 38 degrees Celsius)
* inability to complete FACES pain scale
* evidence of acute chest syndrome clinically or radiographically
* deemed by attending physician to be so ill as to need immediate hospital admission.

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2012-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renee Quarrie, MD, Principal Investigator — Nationwide Childrens Hospital

REFERENCES:
- [Background] Raphael JL, Mei M, Mueller BU, Giordano T. High resource hospitalizations among children with vaso-occlusive crises in sickle cell disease. Pediatr Blood Cancer. 2012 Apr;58(4):584-90. doi: 10.1002/pbc.23181. Epub 2011 May 16. PMID 21584938
- [Background] Mousa SA, Al Momen A, Al Sayegh F, Al Jaouni S, Nasrullah Z, Al Saeed H, Alabdullatif A, Al Sayegh M, Al Zahrani H, Hegazi M, Al Mohamadi A, Alsulaiman A, Omer A, Al Kindi S, Tarawa A, Al Othman F, Qari M. Management of painful vaso-occlusive crisis of sickle-cell anemia: consensus opinion. Clin Appl Thromb Hemost. 2010 Aug;16(4):365-76. doi: 10.1177/1076029609352661. Epub 2010 Jun 7. PMID 20530056
- [Background] Raphael JL, Kamdar A, Wang T, Liu H, Mahoney DH, Mueller BU. Day hospital versus inpatient management of uncomplicated vaso-occlusive crises in children with sickle cell disease. Pediatr Blood Cancer. 2008 Sep;51(3):398-401. doi: 10.1002/pbc.21537. PMID 18300322
- [Background] Raphael JL, Kamdar A, Beavers MB, Mahoney DH, Mueller BU. Treatment of uncomplicated vaso-occlusive crises in children with sickle cell disease in a day hospital. Pediatr Blood Cancer. 2008 Jul;51(1):82-5. doi: 10.1002/pbc.21483. PMID 18383165
- [Background] Field JJ, Knight-Perry JE, Debaun MR. Acute pain in children and adults with sickle cell disease: management in the absence of evidence-based guidelines. Curr Opin Hematol. 2009 May;16(3):173-8. doi: 10.1097/MOH.0b013e328329e167. PMID 19295432
- [Background] Mehta SR, Afenyi-Annan A, Byrns PJ, Lottenberg R. Opportunities to improve outcomes in sickle cell disease. Am Fam Physician. 2006 Jul 15;74(2):303-10. PMID 16883928
- [Background] Platt OS, Thorington BD, Brambilla DJ, Milner PF, Rosse WF, Vichinsky E, Kinney TR. Pain in sickle cell disease. Rates and risk factors. N Engl J Med. 1991 Jul 4;325(1):11-6. doi: 10.1056/NEJM199107043250103. PMID 1710777
- [Background] Conran N, Franco-Penteado CF, Costa FF. Newer aspects of the pathophysiology of sickle cell disease vaso-occlusion. Hemoglobin. 2009;33(1):1-16. doi: 10.1080/03630260802625709. PMID 19205968
- [Background] Jaja SI, Gbadamosi TA, Kehinde MO, Gbenebitse S. The effect of warmth or/and vitamin E supplementation on forearm blood flow and forearm vascular resistance in sickle cell and non sickle cell anaemia subjects. Niger Postgrad Med J. 2003 Mar;10(1):6-12. PMID 12717457

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Warm Fluid | Room Temperature Fluid
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Warm Fluid | Room Temperature Fluid | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.3 (4.7) | 13.6 (5.6) | 14 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 23 | 42
  Male | 21 | 17 | 38
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Rate of Hospital Admission
Description: After being treated for pain in the Emergency Department, the disposition of the patient (whether admitted to the hospital for further care or discharge to home) was recorded.
Time Frame: 4 hours
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Warm Fluid | Room Temperature Fluid
Number analyzed (Participants) | 40 | 40
percentage of participants | 63 [48 to 78] | 55 [40 to 70]

2. Secondary Outcome: Difference in Pain Score
Description: During the ED stay, patient's pain scores on the Wong-Baker FACES scale was recorded at 30 minute intervals until disposition decided. The difference between the pain score upon arrival and at discharge was assessed. Minimum value 1, maximum value 10 (most pain)
Time Frame: 4 hours
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Warm Fluid | Room Temperature Fluid
Number analyzed (Participants) | 40 | 40
units on a scale | -2.6 (3.5) | -2.9 (3.4)

3. Secondary Outcome: Time to Disposition
Description: The amount of time spent in the ED was recorded for each patient
Time Frame: 4 hours
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Warm Fluid | Room Temperature Fluid
Number analyzed (Participants) | 40 | 40
minutes | 158 [140 to 175] | 155 [135 to 175]

4. Secondary Outcome: Amount of Narcotic Administered
Description: The amount of opioid analgesic administered in the ED prior to disposition was recorded for each patient
Time Frame: 4 hours
Measure: Mean (95% Confidence Interval); unit: mg/kg
Arm/Group | Warm Fluid | Room Temperature Fluid
Number analyzed (Participants) | 40 | 40
mg/kg | 0.31 [0.23 to 0.39] | 0.3 [0.23 to 0.38]

5. Secondary Outcome: Global Comfort
Description: Upon disposition patients were asked to complete a survey which assessed their global comfort during the ED stay. Question 2 of the survey addressed comfort by asking: "On a scale of 1 to 5, how do you think the fluid made you feel?" (1 is worse and 5 is better).
Time Frame: 4 hours
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Warm Fluid | Room Temperature Fluid
Number analyzed (Participants) | 29 | 27
units on a scale | 4 [3 to 4] | 3 [3 to 5]

ADVERSE EVENTS:
Arm/Group | Warm Fluid | Room Temperature Fluid
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes